CLINICAL TRIAL: NCT06053892
Title: Comparison of Time for Prucedure, and Effectiveness Between Augmented Reality Enhanced Ultrasound-guided Versus Standard Ultrasound or Fluoroscopic Injections
Brief Title: AR US Versus sUS or Fluoroscopic Injections for Shoulder Punction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting and implementing the study design due to missing ressources.
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R471
Record Dates: First submitted 2023-05-15; First posted 2023-09-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Ultrasound; Interventions

STUDY DESIGN:
Masking Description: The assignment into the study groups is going to be performed by 1:1 randomization using randomisation cards which are drawn by author-ised study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AR US (Active Comparator): Augmented reality sonography guidance for shoulder punctures
  Interventions: Diagnostic Test: Puncture
- standard US (Active Comparator): standard sonography guidance for shoulder punctures
  Interventions: Diagnostic Test: Puncture
- Fluoroscopic (Active Comparator): Fluroscopic guidance for shoulder punctures
  Interventions: Diagnostic Test: Puncture

INTERVENTIONS:
Diagnostic Test: Puncture — Shoulder puncture with the newly designed technique using AR to overlie the US image to the imaged anatomical structures in comparision to standard US and flurosopic-guidance.

SUMMARY:
The goal of this clinical trial is to prospectively evaluate the potential benefits of injections with Augmented Reality enhanced Ulrasound versus standard Ultrasound or fluoroscopy participants where assigend for fluoroscopic joint injections oder for Ultrasound guided injection.

The main question[s] it aims to answer are:

* The primary objective is to evaluate the duration of the different interventions
* the count of needle passes
* assess the reduction of radiation exposure using AR US rather than fluoroscopic guidance for joint injections

DETAILED DESCRIPTION:
Patients assigned for standard Ultrasound or fluoroscopic joint injection are informed about the trial. Participants are randomly assigned to the study or control intervention. 1:1 randomization is used.

In both groups, data on duration of the intervention, count of needle passes, correctness of injection location and radiation exposure will be collected. The outcome measures will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* - Patients 18 to 99 years of age
* Patients assigned for fluoroscopic guided injections (including MR arthrographies)
* Patients assigned for US guided injections (including MR arthrographies)

Exclusion Criteria:

* - Patients who are not willing to be part of the study
* Contraindication against fluoroscopic guided injection
* Women who are pregnant or breast feeding (Pregnancy assessment is part of the routine prior to fluoroscopic joint injections. No pregnancy test will be done for this study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Augmented reality sonography is less time consuming | 10 minutes
  Puncturing shoulders with Augmented reality sonography is faster (measuring the time in minutes and seconds) than when using standard sonography- from point of entry the skin until the target

SECONDARY OUTCOMES:
Sonography is more efficient than fluoroscopic- guidance in shoulder puncturing | 10 minutes (ml aspirated) to 3 days (laboratory results)
  More fluid (measured in ml) can be aspirated with lower false negative results (laboratory results) when puncutring shoulders with US-guidance in comparison to fluoroscopic guidance

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No